CLINICAL TRIAL: NCT05874778
Title: A Multicenter, Phase 2 Study Evaluating the Value of Radiotherapy in Advanced Diffuse Large B-cell Lymphoma Patients With Extranodal Involvement and Large Tumors Who Had Complete Remission as Assessed by PET-CT After Immune-chemotherapy
Brief Title: A Multicenter, Phase 2 Study Evaluating the Value of Radiotherapy in Advanced Diffuse Large B-cell Lymphoma Patients With Extranodal Involvement and Large Tumors Undergoing Immunochemotherapy for PET-CT Assessment of Complete Remission
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023NHLRT01
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Advanced Diffuse Large B-Cell Lymphoma; Extra-nodal Involvement, Large Mass; Radiotherapy
Keywords: Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation Group (Experimental): Paients will be treated with 6-8 cycles (21 days per cycle) of standard R-CHOP chemotherapy.
  After completing the standard immunochemotherapy, subjects will be randomly divided into the radiotherapy group or the non-radiotherapy group, and the curative effects will be evaluated every three months after the end of the treatment or after a patient's leaving the group, so as to obtain the relevant data including those for figuring up 2-year PFS and survival of subjects and any treatment-related side effects as well.
  Interventions: Drug: 6-8 cycles (21 days per cycle) of Standard R-CHOP chemotherapy; Radiation: Radiotherapy beyond standard R-CHOP Chemotherapy
- Non-radiation Group (Active Comparator): Paients will be treated with 6-8 cycles (21 days per cycle) of standard R-CHOP chemotherapy, but after this treatment patients will not be further given radiation therapy.
  Interventions: Drug: 6-8 cycles (21 days per cycle) of Standard R-CHOP chemotherapy

INTERVENTIONS:
Drug: 6-8 cycles (21 days per cycle) of Standard R-CHOP chemotherapy — All enrolled patients will first complete a total of 6-8 cycles (21 days per cycle) of Standard R-CHOP chemotherapy (Rituximab + Cyclophosphamide + Doxorubicin + Prednisolone) and conduct evaluation about treatment effects (i.e. efficacy evaluation) once every 2 cycles, and after their completion of the 6th cycle, they will receive maintenance treatment . After the end of 6th cycle of treatment or after their leaving the group, efficacy evaluation is conducted every three months to obtain relevant data regarding the 2-year Progression-Free Survival(PFS) and survival of the subjects.
Radiation: Radiotherapy beyond standard R-CHOP Chemotherapy — Radiotherapy: after completion of the standard R-CHOP treatment, enrolled patients will be divided into radiotherapy group and non-radiotherapy group. In radiotherapy group, further consolidation radiotherapy targeting patients' pre-treatment large masses or extranodal affected areas will be given, with routine segmentation of 30-36Gy/15-18f.
  Arms: Radiation Group

SUMMARY:
This study is a prospective, single center, phase II clinical study involving 108 patients with primary and late stage Diffuse Large B-cell Lymphoma complicated by large masses and extranodal involvement. The study aims to evaluate the efficacy of radiotherapy targeting large masses and extranodal involvement in treatment-naïve advanced DLBCL patients with large mass lesions and/or extranodal involvement after they had initially been treated with standard immunochemotherapy and received complete remission as assessed by PET-CT.

After completing the standard immunochemotherapy, subjects will be randomly divided into the radiotherapy group or the non-radiotherapy group, and the curative effects will be evaluated every three months after the end of the treatment or after their leaving the group, so as to obtain the relevant data and data of the 2-year Progression Free Survival, survival of the subjects and Treatment-related side effects.

DETAILED DESCRIPTION:
Safety analysis:

The safety analysis is mainly based on descriptive statistical analysis, which lists and describes the incidence, severity, correlation, risk and outcome of adverse events (AE) in this trial.

Efficacy analysis:

The Kaplan-Meier method will be used to draw the overall survival curve and the progression-free survival curve, and to estimate the median survival time, median progression-free survival period and their 95% confidence intervals.

Before starting the study, patients must read and sign the current version of informed consent form approved by the Ethics Committee (EC). All research steps must be carried out within the time window specified in the research schedule.

The duration of safety data collection is from the patient signing the Informed Consent Form (ICF) to the end of the study, with all AEs recorded in the CRF.

The severity of AE will be evaluated based on the NCI CTCAE 5.0 standard. Each patient will undergo a series of planned visits and specific data will be recorded at different time points during the scheduled visits. All examinations/tests are recommended, and the exact examination/test items to be completed during the study shall be subject to clinical practice.

Investigators must be physicians who have been trained in terms of knowledge and conduct of clinical trials and work under the guidance of senior professionals; Prior to the start of the trial, the clinical ward must be inspected so as to ensure its compliance with standardized requirements and to ensure complete readiness of rescue equipment. It is recommended that professional nursing staff administer medication to the subjects and have a detailed understanding of the medication usage to ensure patient compliance; Each investigation site must strictly follow the study protocol; All participating sites should adhere to the ICH-GCP regulations and standard operating procedures (SOPs) for preservation, and all clinical trial information should be recorded, disposed of, and saved for purposes of accurate reporting, interpretation, and verification of study results; Confirm that all data records and reports are correct and complete, and save the original and essential documents related to the study.

This clinical study will be conducted in accordance with the principles established by the 18th World Federation of Medical Associations (Helsinki, 1964) and all subsequent revisions. Before enrollment, it is necessary to weigh the foreseeable risks and inconveniences that study may bring to the subjects against the potential benefits for enrolled patients. Clinical trials can only be initiated and continued when the expected benefits outweigh the risks. Prior to participating in clinical trials, each subject should provide voluntary informed consent, otherwise they cannot be screened or selected.

ELIGIBILITY:
Inclusion Criteria:

1. Using the World Health Organization (WHO) classification of diseases, newly diagnosed diffuse large B-cell lymphoma with large masses (tumor diameter ≥ 7.5cm) and or extranodal involvement patients diagnosed by histology
2. Age: no limit, male or female;
3. ECOG score: 0-2
4. The laboratory meets the following requirements:

   4.1 The bone marrow hematopoietic function is basically normal: WBC ≥ 3.5×10^9/L, ANC ≥ 1.0×10^9/L, PLT ≥ 75 ×10^9/L, Hb ≥ 80g/L;

   4.2 Liver function: AST/ALT≤2×ULN, TBILI≤2×ULN;

   4.3 Renal Function : creatinine clearance rate(Ccr) ≥50ml/min
5. Non-menopausal or non-surgical sterilization female patients of childbearing age must have a serum pregnancy test within 3 days before the first medication, and the result is negative; and they must be non-lactating. Female patients of childbearing age or male patients whose partners are women of childbearing age must agree to use highly effective methods of contraception during the study and within 6 months after the last administration of the study drug;
6. Expected survival period ≥ 6 months;
7. The patient voluntarily joined the study and signed the informed consent;

Exclusion Criteria:

1. Serum pregnancy test positive or breastfeeding women;
2. Lymphoma patients with central nervous system (CNS) invasion;
3. Clinically significant heart disease, including unstable angina, acute myocardial infarction 6 months before randomization, congestive heart failure (NYHA), cardiac function class III or IV; or cardiac left ventricular ejection fraction <50%;
4. Patients with ≥2 grade neuropathy;
5. Patients with active hepatitis B (HBV), hepatitis C (HCV), and other acquired and congenital immunodeficiency diseases;
6. Patients with severe active infection who require systemic antibiotic treatment;
7. Have a history of serious neurological or psychiatric diseases, unable to participate in the trial normally, including dementia, epilepsy, severe depression and mania, etc.;
8. Drug abuse, medical, psychological or social conditions that may interfere with the subject's participation in the research or the evaluation of the research results;
9. Patients considered by the investigator to be unsuitable for enrollment;

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
2-Year Event Free Survival Rate | 2-Year
  The proportion of enrolled patients who are free of events such as death, disease progression, switch to chemotherapy, addition of other treatments, occurrence of fatal or intolerable side effects, and other events
2-Year Progression-Free Survival Rate | 2-Year
  The percentage of people who did not have new tumor growth or cancer spread during or after treatment.

SECONDARY OUTCOMES:
2-Year Overall Survival | 2-Year
  The percentage of enrolled patients who are alive 2 years after their enrollment .
Adverse Events related to Radiotherapy | Adverse events that occur within 30 days
  The occurrence of Hematological and non-Hematological adverse event( NCI CTCAE v5.0）
2-Year Local Control Rate | 2-Year
  The percentage of enrolled patients in radiotherapy group whose tumor volume is equal to or less than their tumor volume at start of radiotherapy